CLINICAL TRIAL: NCT05640440
Title: Executive Function Performance in Children Who Stutter
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Rasha Mohamed Hashem, Assistant lecturer, Sohag University
Other Study IDs: Soh-med-22-11-11
Record Dates: First submitted 2022-11-16; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Stuttering, Childhood; Executive Dysfunction
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children who stutter: assessment executive function and stuttering severity in 30 child with stuttering
  Interventions: Diagnostic Test: Executive function testing
- children who don't stutter: assessment executive function in 30 child with stuttering
  Interventions: Diagnostic Test: Executive function testing

INTERVENTIONS:
Diagnostic Test: Executive function testing — Assessment of executive function subdivision

SUMMARY:
The study aims to asses the executive function in children who stutter for better management of those children

DETAILED DESCRIPTION:
It is a case control study which will be done on 30 child who stutter and 15 normal child as a control group. Executive function testing will be done using computerized program called PEPL . Also, total intelligence quation(IQ) , verbal IQ, non verbal IQ will be assessed in both groups. stuttering severity will be assessed in case group.

ELIGIBILITY:
Inclusion Criteria:

1. Patient and volunteers age between 7 years and 15 years.
2. IQ ≥ 85.

Exclusion Criteria:

* History of secondary stuttering.
* Language impairment and other speech problem.
* Concurrent or history of psychiatric, cognitive, neurological disorders or hearing impairment.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 30 case group, 15 control group age range 7 yrs old and 15 yrs old
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
PEPL numerical stroop test | one year
  Using the Psychological Experimental Building Language (PEBL) current version 2.1 released at 2018 (Muller & Piper, 2014). The test measuring inhibitory function It asses the reaction time in seconds, the total numbers of errors ranging between 0-200
Cognitive flexibility function (sub-division of executive function testing) | one year
  PEPL Berg's Card Sorting Test 64 version of Berg's (1948) Wisconsin Card Sorting Test. The child is asked to sort multi-attribute cards into piles according to an unknown and changing rule. It provides an indication of which rule (shape, color or number) is easiest for the individual. It aims to asses Number of Correct Responses: ranging between 0-64 Number of Total Errors ranging between 0-64 Percent of Perseverative Responses Percent of Perseverative Errors Percent of Non-Perseverative Errors Number of Unique Errors
Working memory score | one year
  Sub-test of Stanford-Binet Intelligence Scales, 5th Edition (SB5) The score ranging between 40-130

SECONDARY OUTCOMES:
Non word Repetation score(Fawzy et al., 2012) | one year
  To test the working memory abilities. the child is asked to repeat a number of non sense words. The score ranges between 0 to 30
Backward digit span score (Aboras et al., 2008) | one year
  It test the working memory. The child is asked to retell a number of digit in backward manner. The score ranges between 0 to 14.

CONTACTS AND LOCATIONS:
Overall Officials: Ahlam A Nabieh, professor, Study Director — ahlaama@yahoo.com
Locations (1):
- Rasha Mohamed Hashem, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided